CLINICAL TRIAL: NCT02453529
Title: A Phase 1, Multiple-Dose, Open-Label Study to Determine and Compare Plasma and Intrapulmonary Concentrations of WCK 4873 in Healthy Adult Human Subjects
Brief Title: Study to Determine and Compare Plasma and Intrapulmonary Concentrations of WCK 4873 in Healthy Adult Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: W-4873-101
Record Dates: First submitted 2015-04-17; First posted 2015-05-25 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: plasma concentration; pulmonary concentration
MeSH Terms: interventions — nafithromycin

ARMS (1):
- WCK 4873 (Experimental): Oral tablets
  Interventions: Drug: WCK 4873

INTERVENTIONS:
Drug: WCK 4873 — Oral tablets

SUMMARY:
This is a Phase 1, multiple dose, open-label pharmacokinetic study conducted in healthy adult male and female subjects.

Subjects will receive 3 oral doses of WCK 4873 administered once-daily starting on Day 1. Blood collection for determining plasma WCK 4873 concentrations will be conducted within 15 minutes prior to and at 1, 2, 3, 4, 6, 9, 12, and 24 hours after the first dose of WCK 4873. The 24 hours post-dose sample after the first dose will be collected prior to Day 2 dosing. Blood samples for determining plasma WCK 4873 concentrations will also be collected within 15 minutes prior to and at 1, 2, 3, 4, 6, 9, 12, 24 and 36 hours after the third dose. Each subject will undergo one standardized bronchoscopy with bronchoalveolar lavage (BAL) in the outpatient bronchoscopy suite at 3, 6, 9, 12, 24 or 48 hours after the third oral dose of WCK 4873. Subjects scheduled for bronchoscopy at 48 hours will also have blood sample drawn for determining plasma WCK 4873 concentrations at 48 hours after the third dose.

Safety will be assessed throughout the study by adverse event monitoring, clinical laboratory tests (including liver function tests), ECG, physical examination and vital sign monitoring. Subjects will discontinue study drug administration in the event of AST/ALT elevation of greater than 3 times the upper limit of normal.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.5 and 30 (kg/m2) and weight between 55.0 and 100.0 kg (both inclusive).
* Medical history without any major pathology as judged by the Principal Investigator.
* Resting supine blood pressure 100-139 (systolic) or 60-89 (diastolic) mm Hg, a resting pulse rate of 40 beats per minute or higher, and showing no clinically relevant deviations as judged by the Principal Investigator.

Exclusion Criteria:

* History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Positive alcohol breath test or urine drug screen test at screening or confinement.
* Positive testing for HIV, Hepatitis B or Hepatitis C.
* Clinically significant pulmonary or any other disease that prevents a subject from undergoing bronchoscopy with pulmonary lavage.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
• Epithelial lining fluid (ELF) and alveolar macrophage (AM) will be used to assess the concentrations of oral WCK 4873 in healthy adult subjects | 48 hrs per dose

SECONDARY OUTCOMES:
• Safety and tolerability of oral WCK 4873 in healthy adult subjects as measure by safety lab assesments, ECGs, physical examinations and AEs captured. | 8 weeks
• Pharmacokinetic (PK) profile of multiple doses (800 mg) of WCK 4873 in healthy adult subjects | 48 hrs last dose
  Plasma concentrations of WCK 4873; plasma PK parameters (Cmax, tmax, kel, t½, AUC0-t, AUC0-24, Vd, CL); ELF concentrations of WCK 4873; concentration of WCK 4873 in alveolar macrophages

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates, 1112 E. McDowell Rd., Phoenix, Arizona, United States

REFERENCES:
- [Derived] Rodvold KA, Gotfried MH, Chugh R, Gupta M, Friedland HD, Bhatia A. Comparison of Plasma and Intrapulmonary Concentrations of Nafithromycin (WCK 4873) in Healthy Adult Subjects. Antimicrob Agents Chemother. 2017 Aug 24;61(9):e01096-17. doi: 10.1128/AAC.01096-17. Print 2017 Sep. PMID 28696231